CLINICAL TRIAL: NCT06846216
Title: Evaluation of the Combined Application of BTL-785F and HPM-6000UF Devices for Women's Intimate Wellness
Brief Title: Combination of BTL-785F and HPM-6000UF Devices for Women's Intimate Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS700
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Vulvovaginal Atrophy; Urinary Incontinence; Sexual Dysfunction
Keywords: vulvovaginal atrophy; urinary incontinence; sexual dysfunction; radiofrequency; HIFEM; urogenital system
MeSH Terms: conditions — Urinary Incontinence; Sexual Dysfunction, Physiological | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-785F and HPM-6000UF Devices (Experimental): Subjects will undergo six treatment sessions.
  Interventions: Device: Treatment with BTL-785F and HPM-6000UF Devices

INTERVENTIONS:
Device: Treatment with BTL-785F and HPM-6000UF Devices — Three treatment sessions will consist of the consecutive application of the BTL-785F and HPM-6000UF devices, delivered 5-10 days apart. Three sessions will consist of the standalone application of the HPM-6000UF device, delivered 2-4 days apart. The treatments with BTL-785 device equipped with BTL-785-3 applicator will last 2-10 minutes and with HPM-6000UF 28 minutes.

SUMMARY:
The goal of this clinical trial is to evaluate the combined application of BTL-785F and HPM-6000UF Devices in improving quality of life in women with negative changes in the urogenital system (vulvovaginal atrophy symptoms, urinary incontinence or sexual dysfunction). The main question it aims to answer is:

Does the combined application of BTL-785F and HPM-6000UF Devices reduces the score of the Vulvovaginal Symptoms Questionnaire?

Participants will:

* Undergo 6 treatment sessions.Three sessions will consist of combined application of BTL-785F and HPM-6000UF devices and three sessions will consist of standalone application of the HPM-6000UF device.
* Attend follow-up visits
* Complete questionnaires

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and performance of the combined application of the BTL-785F and HPM-6000UF devices for the improvement of Quality of Life in Women with in the urogenital system (vulvovaginal atrophy symptoms, urinary incontinence or sexual dysfunction). This clinical trial uses a multicenter, single-arm, open-label, interventional design. Subjects will undergo six treatment sessions.

Follow-up visits are scheduled 1 month, 3 months, and 6 months after the last treatment session.

Participants will complete the Vulvovaginal Symptoms Questionnaire, King's Health Questionnaire, and the 6-item Female Sexual Function Questionnaire, which will be administered at the baseline visit, after the last treatment, and all follow-up visits. Additionally, the Subject Satisfaction Questionnaire, given after the last treatment and at all follow-up visits, will be filled out. Therapy Comfort Questionnaire will be administered after the last treatment. During the study duration, observation for adverse events and side effects will take place.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects aged 30 years or older seeking treatment for intimate concerns such as negative changes in the vulvovaginal area, impairment of sexual function, and UI.
* The subject has had at least one full-term pregnancy with vaginal delivery or a C-section.
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits, and side effects, and must sign the Informed Consent Form.
* The subject is willing and able to abstain from partaking in any concurrent treatments of aggravating vulvovaginal changes, other than the study procedures during study participation.
* Willingness to comply with study instructions and to return to the clinic for the required visits.
* Women of childbearing potential are required to use birth control measures.

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants including Intrauterine metal devices
* Nuvaring (Birth Control Vaginal Ring)
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before - complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitivity disorders in the treatment area
* Varicose veins, pronounced edemas
* Sexually transmitted infection
* Pelvic organ prolapsed beyond the hymenal ring and evidence of fine rectovaginal septum
* Undergoing pelvic floor physiotherapy
* Implanted neurostimulators
* Pulmonary insufficiency
* Drug pumps
* Malignant tumor
* Increased body temperature (above 99°F) and fever (above 100.4 °F)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Quality of Life of Women with Vulvovaginal Atrophy Symptoms | 12 months
  The change in the score obtained from the Vulvovaginal Symptoms Questionnaire will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, and at the 1-month, 3-month, and 6-month follow-up visits. The score ranges from 0 to 16 for sexually inactive women and from 0 to 20 for sexually active women. An improvement is defined as a decrease in score.

SECONDARY OUTCOMES:
Assessment of Change in Quality of Life of Women with Urinary Incontinence | 12 months
  The change in the score obtained from the King's Health Questionnaire will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, and at the 1-month, 3-month, and 6-month follow-up visits. The score ranges between 0 to 100 for the nine domains, and between 0 to 30 for the Symptom Severity Scale. An improvement is defined as a decrease in score.
Assessment of Change in Sexual Functioning | 12 months
  The change in the score obtained from the 6-item Female Sexual Function Index will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, and at the 1-month, 3-month, and 6-month follow-up visits. The score ranges between 0 to 30. An improvement is defined as an increase in score.
Assessment of Therapy Comfort | 12 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Pain Rating Scale (0 = no pain, 10 = worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Pain Rating Scale indicate higher therapy comfort.
Assessment of Satisfaction | 12 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Subject Satisfaction questionnaire. The questionnaire will be administered after the last treatment, and at the 1-month, 3-month, and 6-month follow-up visits. Responses to questions about the treated urogenital area will range from "strongly agree" (1 point) to "strongly disagree" (5 points). A higher score for each statement indicate better outcomes.
Incidence of Treatment-related Adverse Events | 12 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the combined application of the BTL-785F and HPM-6000UF devices and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Pelvic Health and Wellness, Mission Viejo, California
  - Kimberly L. Evans MD, PLLC, Sugar Land, Texas